CLINICAL TRIAL: NCT04761120
Title: Annuloplasty Rings and Band Post-Market Clinical Follow-Up (ARB-PMCF) Study
Brief Title: Annuloplasty Rings and Band Post-Market Clinical Follow-Up Study
Acronym: ARB-PMCF
Status: Recruiting | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: ABT-CIP-10368
Record Dates: First submitted 2021-02-12; First posted 2021-02-18 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-02

CONDITIONS: Mitral Regurgitation; Tricuspid Regurgitation; Valvular Heart Disease
Keywords: Mitral Regurgitation; Tricuspid Regurgitation; Valve Surgery; Valve Repair; Annuloplasty Rings; Annuloplasty Bands; Rigid Saddle Ring; Séguin Annuloplasty Ring; Tailor Annuloplasty Ring; Tailor Annuloplasty Band
MeSH Terms: conditions — Mitral Valve Insufficiency; Tricuspid Valve Insufficiency; Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (5):
- Group 1: Primary mitral disease repair surgery with an Abbott annuloplasty ring implant: Group 1 will enroll 200 subjects undergoing surgical repair of primary mitral regurgitation that includes annuloplasty with an Abbott SJM Rigid Saddle Ring, Séguin Ring or full Tailor Ring without cut zone removal. Enrollment must include at least 50 subjects implanted with each ring model. In primary mitral regurgitation, backflow through the closed valve is caused by disease intrinsic to the mitral valve tissue itself.
  Interventions: Device: Abbott SJM Rigid Saddle Ring; Device: Abbott SJM Séguin Ring; Device: Abbott SJM Tailor Ring
- Group 2: Secondary mitral disease repair surgery with an Abbott annuloplasty ring implant: Group 2 will enroll 200 subjects undergoing surgical repair of secondary mitral regurgitation that includes annuloplasty with an Abbott SJM Rigid Saddle Ring, Séguin Ring or full Tailor Ring without cut zone removal. Enrollment must include at least 50 subjects implanted with each ring model. In secondary mitral regurgitation, backflow through the closed valve is secondary to diseases of the surrounding myocardium, rather than caused by disease of the valve tissue itself.
  Interventions: Device: Abbott SJM Rigid Saddle Ring; Device: Abbott SJM Séguin Ring; Device: Abbott SJM Tailor Ring
- Group 3: Primary tricuspid disease repair surgery with a full Tailor Ring implant: Group 3 will enroll up to 50 subjects undergoing surgical repair of primary tricuspid regurgitation that includes annuloplasty with a full Abbott SJM Tailor Ring without cut zone removal. In primary tricuspid regurgitation, backflow through the closed valve is caused by disease intrinsic to the tricuspid valve tissue itself.
  Interventions: Device: Abbott SJM Tailor Ring
- Group 4: Secondary tricuspid disease repair surgery with a full Tailor Ring implant: Group 4 will enroll up to 50 subjects undergoing surgical repair of secondary tricuspid regurgitation that includes annuloplasty with a full Abbott SJM Tailor Ring without cut zone removal. In secondary tricuspid regurgitation, backflow through the closed valve is secondary to diseases of the surrounding myocardium, rather than caused by disease of the valve tissue itself.
  Interventions: Device: Abbott SJM Tailor Ring
- Group 5: Primary tricuspid disease repair surgery with a partial Tailor Ring or Tailor Band implant: Group 4 will enroll up to 50 subjects undergoing surgical repair of secondary tricuspid regurgitation that includes posterior annuloplasty with either a partial Abbott SJM Tailor Ring with cut zone removed or an Abbott SJM Tailor Band. In primary tricuspid regurgitation, backflow through the closed valve is caused by disease intrinsic to the tricuspid valve tissue itself.
  Interventions: Device: Abbott SJM Tailor Ring; Device: Abbott SJM Tailor Band

INTERVENTIONS:
Device: Abbott SJM Rigid Saddle Ring — The Abbott SJM Rigid Saddle Ring is a rigid, polyester-velour-covered, titanium alloy mitral annuloplasty ring with a saddle shape intended to mimic the shape of a healthy mitral annulus during systole.
  Groups: Group 1: Primary mitral disease repair surgery with an Abbott annuloplasty ring implant; Group 2: Secondary mitral disease repair surgery with an Abbott annuloplasty ring implant
Device: Abbott SJM Séguin Ring — The Abbott SJM Séguin Ring is a semi-rigid, polyester-velour-covered, polyethylene mitral annuloplasty ring that varies in thickness and flexibility over its circumference, with the posterior portion of the ring having greater flexibility than the anterior portion.
  Groups: Group 1: Primary mitral disease repair surgery with an Abbott annuloplasty ring implant; Group 2: Secondary mitral disease repair surgery with an Abbott annuloplasty ring implant
Device: Abbott SJM Tailor Ring — The Abbott SJM Tailor Ring is a flexible, polyester-velour-covered, silicone annuloplasty ring indicated for use in surgical repair of the mitral or tricuspid valve. The Tailor Ring can be implanted as a full annuloplasty ring, or the surgeon can remove the ring's cut zone with a scalpel and use the partial Tailor Ring as a posterior annuloplasty band.
Device: Abbott SJM Tailor Band — The Abbott SJM Tailor Band is a flexible, polyester-velour-covered, silicone band for posterior annuloplasty indicated for use in surgical repair of mitral or tricuspid valve. The Tailor Band is identical to the Tailor Ring with the cut zone removed, save that the polyester covering is sewn closed at the ends of the band during manufacturing.
  Groups: Group 5: Primary tricuspid disease repair surgery with a partial Tailor Ring or Tailor Band implant

SUMMARY:
ARB-PMCF is a multicenter, observational study of the safety and performance of Abbott annuloplasty devices used in surgical repair of mitral and tricuspid valve regurgitation. The devices included in this study are the SJM™ Rigid Saddle Ring and SJM Séguin Annuloplasty Ring, indicated for mitral valve repair, and the SJM Tailor™ Annuloplasty Ring and SJM Tailor Annuloplasty Band, indicated for mitral or tricuspid repair. Participants will be enrolled prior to undergoing mitral or tricuspid valve repair surgery including an Abbott annuloplasty implant and will complete annual follow-up visits through five years from implant. The study is being conducted to meet post-market clinical follow-up requirements of the European Union Medical Device Directives.

DETAILED DESCRIPTION:
The ARB-PMCF Study has a prospective, multicenter, observational, parallel group design in which up to 550 subjects will be followed through five years from implant of an Abbott annuloplasty device, with or without concomitant procedures, in five treatment groups, including primary mitral disease repair (N=200) with the Rigid Saddle Ring, Séguin Ring or full Tailor Ring without cut zone removal; secondary mitral disease repair (N=200) with the Rigid Saddle Ring, Séguin Ring or full Tailor Ring; primary tricuspid disease repair with the full Tailor Ring (N=50); secondary tricuspid disease repair with the full Tailor Ring (N=50); and primary tricuspid disease repair with the Tailor Band or partial Tailor Ring with cut zone removed (N=50). Study enrollment will occur at up to 25 global centers with approximately half or more of all implanted subjects being from European sites. The study will enroll adult subjects expected to be implanted with an Abbott annuloplasty device within 90 days who meet all other eligibility requirements. Participants will complete annual in-clinic or telephone follow-up visits through five years from their annuloplasty implant. Data collected will include adverse events, cardiac medication usage, New York Heart Association functional classification (a measure of the severity of heart failure symptoms) and echocardiographic assessments of regurgitation through the repaired valve.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is expected to undergo cardiac surgery in ≤90 days including at least one of the following:

   1. implant of a Rigid Saddle Ring, Séguin Ring or a full Tailor Ring without cut zone removal for MR repair
   2. implant of a full Tailor Ring without cut zone removal for TR repair, or
   3. implant of a Tailor Band or partial Tailor Ring with cut zone removed for primary TR repair.
2. Subject's cardiac surgery will be performed by a study investigator.
3. Subject will be ≥18 years old at the time of their annuloplasty implant(s).
4. Subject provides written informed consent and agrees to comply with all required study visits and procedures.

Exclusion Criteria:

1. Subject is below the age of legal consent in the applicable jurisdiction or otherwise lacks legal authority to provide informed consent.
2. Subject is unable to read or write or has a mental illness or disability that impairs their ability to provide written informed consent.
3. Subject is expected to have active endocarditis at the time of their Abbott annuloplasty device implant(s).
4. Subject cannot be unambiguously assigned to a treatment group due to missing data on repair indication(s) or the model and configuration (cut zone removed or not) of their Abbott annuloplasty implant(s).
5. Subject is participating in another clinical investigation including any treatment outside the investigative site's usual standard of care.
6. Subject has anomalous anatomy or medical, surgical, psychiatric or social history or conditions that, in the investigator's opinion, would limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll male and female adult subjects from the general population of cardiac surgery patients who are expected to be implanted with a Rigid Saddle, Séguin or full Tailor Ring for mitral regurgitation (MR) repair, a full Tailor Ring for tricuspid regurgitation (TR) repair or a Tailor Band or partial Tailor Ring for primary TR repair within 90 days.
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2030-11 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants in Each Treatment Group with Freedom from All-Cause Mortality through 5 Years Post-Implant | 5 years
  Percentage of participants in each study treatment group (Groups 1 through 5) who are free of death from any cause through 5 years after their Abbott annuloplasty device implant, estimated from time-to-event data using the Kaplan-Meier estimator. This outcome will be reported for each treatment group separately.
Percentage of Participants in Each Mitral Treatment Group with Freedom from Reoperation or Transcatheter Reintervention for Mitral Regurgitation through 5 Years Post-Implant | 5 years
  Percentage of participants in each mitral treatment group (Groups 1 and 2) who are free from reoperation or transcatheter intervention for mitral regurgitation through 5 years after their Abbott annuloplasty implant, estimated from time-to-event data using the Kaplan-Meier estimator. This outcome will be reported separately for Group 1 and Group 2.
Percentage of Participants in Each Tricuspid Treatment Group with at least a 1-Class Reduction in New York Heart Association (NYHA) Functional Classification at 1 Year Post-Implant. | 1 year
  This outcome will be reported for each tricuspid repair group (Groups 3 through 5) separately. NYHA functional classification is a widely used indicator of the severity of heart failure symptoms with four classes:
  Class I. No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, or dyspnea (shortness of breath).
  Class II. Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, or dyspnea.
  Class III. Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea.
  Class IV. Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest. If any physical activity is undertaken, discomfort increases.

SECONDARY OUTCOMES:
Number of Participants in Each Treatment Group by Grade of Regurgitation in the Valve Undergoing Repair, Pre-Operatively, at Discharge, and at 1, 3 and 5 Years Post-Implant | Pre-Operative Baseline, within 60 days post-implant, and 1, 3 and 5 years post-implant
  This outcome will be reported for each treatment group separately at each timepoint. Regurgitation occurs when a heart valve does not fully seal, allowing backflow of blood through the closed valve. Mitral and tricuspid valve regurgitation in this study will be graded as none/trivial, mild, moderate or severe by echocardiographic assessment. Moderate or severe regurgitation can cause symptoms of heart failure, such as fatigue, shortness of breath and exercise intolerance.
Number of Participants in Each Treatment Group by NYHA Functional Class, Pre-Operatively and at Discharge, 1, 3 and 5 Years Post-Implant. | Pre-Operative Baseline, within 60 days post-implant, and 1, 3 and 5 years post-implant
  This outcome will be reported for each treatment group separately at each timepoint. NYHA functional classification is a widely used indicator of the severity of heart failure symptoms with four classes:
  Class I. No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, or dyspnea (shortness of breath).
  Class II. Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, or dyspnea.
  Class III. Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea.
  Class IV. Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest. If any physical activity is undertaken, discomfort increases.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Palmer, Study Director — Abbott
Locations (17):
- United States (2):
  - Duke University Hospital, Durham, North Carolina
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- Tartu University Hospital, Tartu, Estonia
- France (2):
  - Hopital Cardiovasculaire et Pneumologique Louis Pradel, Lyon, Auvergne-Rhône-Alpes
  - CHU de Besançon - Jean Minjoz, Besançon, Bourgogne-Franche-Comté
- Germany (5):
  - Herzchirurgische Abteilung Klinikum Passau, Passau, Bavaria
  - Universitätsklinikum Würzburg, Würzburg, Bavaria
  - Herzzentrum-Bremen Klinikum Links der Weser, Bremen, City state Bremen
  - Herzzentrum Dresden, Universitätsklinik an der Technischen Universität Dresden, Dresden, Saxony
  - Universitätsklinikum Jena, Jena, Thuringia
- Italy (5):
  - Policlinico S.Orsola-Malpighi, Bologna, Bologna
  - Ospedale San Raffaele - Cardiac, Milan, Lombardy
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Lombard
  - Ospedale Luigi Sacco, Milan, Milan
  - Ospedale Umberto I, Turin, Piedmont
- Catharina Ziekenhuis, Eindhoven, North Brabant, Netherlands
- Hospital Alvaro Cunqueiro, Vigo, Pontevedra, Spain

IPD SHARING:
Plan to Share IPD: No